CLINICAL TRIAL: NCT00161057
Title: Functional Brain Activation Patterns in Schizophrenia, Measured Before and After Treatment
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: divisie hersenen, UMC Utrecht
Other Study IDs: METC 01/134
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Schizophrenia; Schizophreniform Disorders
Keywords: Schizophrenia; Medication-naive; Functional MRI; Working memory; Language lateralization; schizoaffective disorder; psychotic disorder Not Otherwise Specified
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In this study we, the investigators at UMC Utrecht, intend to investigate changes in brain activation patterns using functional magnetic resonance imaging (MRI), in patients suffering from schizophrenia who are medication naive or off medication, before using medication and after 8 weeks of medication. Patients will perform a working memory task, a language task and a motor task while lying in the scanner. We hypothesize that the efficiency of the working memory system is reduced and that the lateralization of language is diminished in these patients, and that these functions will normalize after treatment.

DETAILED DESCRIPTION:
Schizophrenia is a heterogeneous disorder with a wide range of symptoms and signs including hallucinations, delusions, disorganisation, negative symptoms and cognitive deficits. Investigation of the neural substrates of the cognitive deficits in schizophrenia has revealed abnormalities in brain activity patterns. Particularly, earlier studies using functional FMRI conducted at the UMCU, revealed diminished language laterality, deficits in working memory and a reduced ability to automate cognitive processes. The aim of this project is to study the relationship between these brain activation patterns and neuroleptic treatment. More insight into psychopharmacological effects on brain physiology, may eventually enable us to better predict what effect treatment will have on patients.

Patients with a confirmed diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder or psychotic disorder not otherwise specified (NOS), who are medication naive or medication free for a period of at least 2 weeks will be included. Patients will be tested before and after 8 weeks of treatment with an atypical antipsychotic. In the scanner patients will perform a working memory task, a language task and a visual-motor task. At study entry and after 8 weeks the PANSS, Clinical Global Impressions (CGI) and CDSS (Calgary Depression Scale of Schizophrenia) will be performed. Besides these patients, we will also include a group of matched healthy controls. We hypothesize that in medication naive or patients of-medication lateralization is reduced, and that efficiency of the working memory system is reduced. Lateralization is expected to correlate negatively with positive functions. We expect that antipsychotic treatment will normalize brain function and that the degree of normalization is correlated with the clinical measures of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria (patients):

* Diagnoses of schizophrenia, schizophreniform disorder, schizoaffective disorder or psychotic disorder NOS, confirmed on the basis of Comprehensive Assessment of Symptoms and History (CASH) or a Structured Clinical Interview for DSM-IV Disorders (SCID) interview
* Ages between 16 and 50 years
* CGI of at least 4
* Patients are neuroleptic-naive or medication-free for at least 2 weeks

Inclusion Criteria (healthy controls):

* No psychiatric disorders (according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition [DSM-IV], Axis I)
* No psychiatric disorders in first degree relatives.
* Ages: between 18 and 50 years old

Exclusion Criteria (patients and healthy controls):

* Ferrous objects in or around the body
* Neurological or medical illness, including closed head injury.
* Mental retardation.
* Diagnosis of substance dependence within the previous 3 months.
* Pregnancy
* Treatment with antidepressants or mood stabilizers within 3 weeks of inclusion.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: first episode schizophrenia patients, medication naive (or medication-free) and matched healthy controls.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2001-12; Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta V Veelen, Principal Investigator — UMC Utrecht; Rene Kahn, M.D. Ph.D., Study Chair — UMC Utrecht
Locations (1):
- Dept. of Psychiatry, UMC Utrecht, Utrecht, Utrecht, Netherlands